CLINICAL TRIAL: NCT05405959
Title: Efficacy of Kinesio Tape Application With Epidermis Dermis Fascia (EDF) Technique in Patients With Active Myofascial Trigger Points in Upper Trapezius Muscle, a Prospective, Double Blinded Sham Controlled Randomized Study
Brief Title: Kinesio Tape Application With EDF Technique on Active Trigger Points of Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Prof, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNEAH-KAEK 2017/109
Record Dates: First submitted 2022-05-26; First posted 2022-06-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Myofascial Pain Syndrome; Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotaping (KT) with EDF technique (Experimental): the patients were seated and asked to flex their neck laterally to the contralateral side and to rotate their head to the same side while the shoulder was adducted. I band was first fold in half and then divided into 5 lines without cutting the ends to form a web shape. Two pieces of web shaped 20-25 cm length KT were used. The end of the KT was applied to the acromion, and the spinal process of C7 vertebra without stretching, but the web on the muscle had %10-15 tension. The second web shaped band was applied using the same technique between acromion and thoracal vertebral insertion of the middle trapezius muscle. Kinesio tape was planned to stay on for five days; it was applied twice, with two days of rest between applications Trapezius stretching exercises were given to patients as home exercise program.
  Interventions: Device: Kinesio tape
- Sham Kinesiotaping (Sham Comparator): The sham group received improper KT application consisting two I strips (same material as the real application) applied with no tension on c7 spinal process as cross sign. For sham taping, the cervical spine of the participants was placed in a neutral position. Kinesio tape was planned to stay on for five days; it was applied twice, with two days of rest between applications Trapezius stretching exercises were given to patients as home exercise program
  Interventions: Device: Sham Kinesio Tape

INTERVENTIONS:
Device: Kinesio tape — The Kinesio Tex Gold FP (Kinesio Tex Tape, Kinesio Holding Corporation, Albuquerque, NM, USA) was used. It was waterproof, porous and adhesive, had a width of 5 cm and a thickness of 0.5 mm. The same brand of tape was used in both groups.
  Arms: Kinesiotaping (KT) with EDF technique
Device: Sham Kinesio Tape — The Kinesio Tex Gold FP (Kinesio Tex Tape, Kinesio Holding Corporation, Albuquerque, NM, USA) was used. It was waterproof, porous and adhesive, had a width of 5 cm and a thickness of 0.5 mm. The same brand of tape was used in both groups.
  Arms: Sham Kinesiotaping

SUMMARY:
In this double-blinded, prospective randomized sham controlled multi centered study, the aim was to investigate the efficacy of EDF technique on pain intensity, number of active TrPs, cervical ROM and disability levels in patients with MPS on upper trapezius (UT) muscle.180 patients were randomly allocated to kinesio taping (KT) group or sham group. Applications were done two times 1 week apart. VAS-pain scores, disability scores , cervical ROM angles and number of trigger points were evaluated as outcome parameters. Vas-pain scores and number of trigger points were assessed at baseline, after 1 week and after 2 weeks (at the end of the study). Cervical ROM angles and disability (measured by Neck Pain Disability Scale) were assessed at baseline and at the end of the study. Both groups received home exercise program. As a result application of KT with EDF technique to the UT muscle provided a significant improvement in pain level, disability, number of active TrPs and cervical ROM angles and found superior to sham application.

DETAILED DESCRIPTION:
In order to determine the sample size, power analysis was performed using the G*Power Version 3.1.9.2 program. Effect size of 1.26 was set up for the VAS pain score changes between groups as per the previous study. For power calculations, a confidence level (α) of 0.05 and a power level of 0.95 was assumed. Fifteen patients per group in each center was required. 15 patients were randomized to two groups in each center by numbered envelopes method. The group 1 and group 2 notes were put into to the closed envelopes separately, and each patient randomly chose an envelope and gave it to a physician who was not the researcher. One researcher evaluated the patient and then collected the data, and the second researcher who was certified as KT practitioner applied the KT. Both patients and the researcher who recorded the data were blinded to treatment allocation.

ELIGIBILITY:
The inclusion criteria:

* presence of an at least one active TrP and palpable taut band in the UT muscle
* pain duration less than 3 months
* pain Visual Analog Score VAS≥4
* being between 18 and 50 years of age

The exclusion criteria:

* diagnosis of neuromuscular, rheumatic, inflammatory diseases
* malignancy
* uncontrollled systemic conditions
* infections
* trauma
* neck surgery
* pregnancy
* obesity (BMI≥ 30 kg/m2).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
pain intensity | Change from baseline at 2nd week
  Visual Analog Scale: The Visual Analog Scale (VAS) (0-10 cm) was used to record each patient's current level of neck pain, with 0 indicating no pain and 10 indicating the worst pain that the patient had experienced.Higher scores mean worse outcome
number of active trigger points | Change from baseline at 2nd week
  number of active trigger points. Trigger points were determined manually by physical examination described by Travell and Simons.
cervical range of motion angles | Change from baseline at 2nd week
  measured by goniometer for flexion, extension, left and right lateral flexion of cervical spine
Disability Level | Change from baseline at 2nd week
  Neck Pain Disability Scale: The questionnaire consists of 20 items and measures neck movements, pain intensity, effect of neck pain on emotion factors, and interference with daily life activities. Each section is scored on a 0-5 rating scale and total score ranges from 0 to 100. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Külcü, prof, Principal Investigator — Haydarpaşa Numune Edutation and Research Hospital; Arzu Dinç, Study Director — Medipol University; Belgin Erhan, Study Chair — Medeniyet University; Birkan Sonel Tur, Study Chair — Ankara University; Gül Tuğba Bulut, Study Chair — Istanbul E%R Hospital; Kamil Yazıcıoğlu, Study Chair — Güven Hospital; Zeynep Alpoğuz, Study Chair — Ankara State Hospital; Elif Çiğdem Keleş, Study Chair — Yeditepe University; Figen Ayhan, Study Chair — Uşak University; Pınar Borman, Study Chair — Hacettepe University; Merve Soysal, Study Chair — Ankara University; Bahar Çakmak, Study Chair — Bakırköy Sadi Konuk Education and Research Hospital
Locations (1):
- Duygu Külcü, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No